CLINICAL TRIAL: NCT05481255
Title: Does the Menstrual Phase Affect Skin Puncture Pain During Spinal Anesthesia? Prospective, Observational Study
Brief Title: Association With Spinal Needle-puncture Pain and Menstrual Phase
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Other Study IDs: spinal needle-puncture pain
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aimed to evaluate the relationship between menstrual phase cycles and spinal needle-puncture pain during spinal anesthesia in female patients of reproductive age.

DETAILED DESCRIPTION:
Before the spinal anesthesia procedure, the anxiety and depression levels of the patients will be evaluated with the 14-scale 'hospital anxiety and depression scale.' The spinal anesthesia procedure will be performed by the anesthesiologist responsible for the patient. At the end of the spinal anesthesia procedure, a researcher with no knowledge of the patient's menstrual phase information will ask rate the spinal needle-puncture pain felt during spinal anesthesia with a numerical rating scale (NRS), which is graded from 1 to 10 (0: no pain, 10: very severe pain).

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers of reproductive age have had a regular menstrual cycle for at least six months

Exclusion Criteria:

* Pregnancy
* ASA physical status III and IV
* Patients with psychiatric disorders,
* Emergency surgeries
* Mentally retarded patients,
* Patients with multiple spinal anesthesia trials
* Patients with previous spinal surgery experience

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only female patients will be involved with regular and active menstrual cycles
Study Population: 80 female patients who are of reproductive age and have had a regular menstrual cycle for at least six months
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
spinal needle-puncture pain | 10 minutes
  A numerical rating scale (NRS) will be used to assess spinal needle-puncture pain during spinal anesthesia, graded from 1 to 10 (0: no pain, 10: very severe pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Education and Training Hospital, Konya, Turkey (Türkiye)